CLINICAL TRIAL: NCT04825379
Title: Clinical Evaluation of a Bioactive Material
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Assoc. Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bioactive-composite
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Tooth Disease
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioactive composite (Experimental): Cention N, Ivoclar Vivadent, Schaan, Liechtenstein (CN)
  Interventions: Device: bioactive composite
- posterior resin composite (Experimental): G-ænial Posterior (GC, Tokyo, Japan) (GP)
  Interventions: Device: posterior composite

INTERVENTIONS:
Device: bioactive composite — Cention N
  Arms: bioactive composite
Device: posterior composite — G-ænial Posterior
  Arms: posterior resin composite

SUMMARY:
The clinical performance of a bioactive composite and a posterior resin composite in class II restorations will be evaluated and compared. After recruiting participants with at least 2 approximal caries lesions, all restorations will be placed by a single clinician. All caries lesions will be removed before restoring. Cavities will be divided into two groups: a bioactive composite [Cention N, Ivoclar Vivadent, Schaan, Liechtenstein (CN)] and a posterior resin composite [G-ænial Posterior (GC, Tokyo, Japan) (GP)] All restorative procedures will be conducted according to manufacturers' instructions. Restorations will be scored using FDI criteria after a week (baseline) 6, 12, 24, 36 and 48 months. Descriptive statistics will be performed using chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* age range will be 18 to 65
* patients should have at least 2 approximal caries lesions require restoration
* healthy periodontal status
* a good likelihood of recall availability

Exclusion Criteria:

* poor gingival health
* adverse medical history
* potential behavioral problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical performances of different restorative systems according to FDI criteria | two years
  Two year results according to FDI criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No